CLINICAL TRIAL: NCT00552734
Title: Glycemic Control and Prevention of Hypoglycemia in Intensively Treated Subjects With Type 1 Diabetes Using Accu-Chek® Advisor Insulin Guidance Software
Brief Title: Improved Glycemic Control in Adult Subjects With Type 1 Diabetes on MDI Using Insulin Guidance Software
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 04-0834
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes
Keywords: Type 1 diabetes; Improved glycemic control; Glucose excursions; Target range glucose levels; Insulin guidance software; Advisor
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: The other half of the patients were randomized to the control group who were followed for their routine diabetes care and had to visit the clinic on the same schedule as the experimental group.
  Interventions: Device: Insulin Guidance Software
- Experimental: Half of the subjects were randomized to this group using insulin guidance software on a PDA to adjust their insulin dose at home based on the prescription provided by the provider.
  Interventions: Device: Insulin Guidance Software

INTERVENTIONS:
Device: Insulin Guidance Software — At baseline a healthcare provider reviewed the features of the software on the PDA and loaded a subject specific insulin dosing algorithm into the software based on the physician's recommendations. The program advised basal, bolus and correction insulin dosages based on individual patients' prescriptions in addition to being alerted for SMBG testing. Subjects in the experimental group were also asked to input their blood glucose values into the PDA via the touch screen. Subjects then received a recommended insulin dose based on their prescription which was programmed by the healthcare provider. The patients were asked to either agree with the recommended insulin dose or disagree, and manually enter the insulin dose they took for a given event.
  Other Names: Accu-Chek Insulin Guidance Software

SUMMARY:
140 subjects will be enrolled into the clinical study and randomized into the Control Group or the Experimental Group by block randomization. The subjects must meet all inclusion and none of the exclusion criteria. Each subject will have 7 clinic visits and 3 phone visits. The Baseline Visit will consist of a complete history, vitals, a physical examination and completion of the consent and screening process. All clinic visits, except for the Baseline Visit will include meter/PDA download. In addition, meter education will be provided to all subjects, and PDA education will be provided to the Experimental group at the Baseline Visit and 2-Week Visit as needed to ensure subject understanding. The phone visits will consist of a history including any changes in insulin dose, and any hypoglycemic events, hyperglycemic events, or other adverse events that have occurred since the last clinic visit.

The primary endpoint in this study was to show a reduction in A1c of at least 0.4% or higher in the insulin guidance software group at 6 months and/or 1 year.

DETAILED DESCRIPTION:
Research Design and Methods A total of 123 adult subjects with type 1 diabetes with a baseline A1c of 7.5-11% were enrolled in the study at the Barbara Davis Center for Childhood Diabetes at the University of Colorado at Denver Health Sciences Center. Two patients screen failed (entry criteria not met) before randomization, leaving 60 subjects randomized to the control group and 61 subjects randomized to the experimental group (Advisor). Subjects were randomized based on lottery system using sealed envelopes. All patients had baseline blood work which included a complete blood count (CBC), complete metabolic panel (CMP), creatnine kinase (CK) and an A1c. The mean A1c at baseline was 8.54 ±0.11 in the control group and 8.42 ±0.11 in the experimental group (p=0.4265).

Subjects were randomized on a 1:1 basis to either the experimental or control group. All subjects in the experimental group received the same training for insulin guidance software program for personal data assistant (PDA). All subjects were given a glucose meter and an unlimited supply of test strips for self monitoring of blood glucose (SMBG). Women who were pregnant or planning to become pregnant were excluded from participation in the study as were patients on insulin pumps, those taking glucocorticoid therapy, and those diagnosed with cancer, liver disease, anemia or hepatitis. Patients who exercised more than five days a week, or often traveled internationally were also excluded.

The protocol was approved by the Colorado Multiple Institutional Review Board (COMIRB). All subjects signed an informed consent form before being enrolled in the study.

Visits All subjects were asked to attend 7 in clinic visits (baseline, 2 week, 6 week, 3 month, 6 month, 9 month and 12 month) and participate in 3 telephone visits (4.5month, 7.5month, 9.5 month) throughout the course of the study. Data for blood glucose values, testing frequency, hyperglycemic excursions, hypoglycemic events (all, nocturnal, and severe), insulin dose, weight and BMI, hospitalizations, emergency room visits and illnesses were recorded at each in clinic visit. All subjects completed a patient satisfaction questionnaire and the experimental group also completed an Advisor questionnaire.

As part of their routine clinical care, any additional phone visits were equally encouraged in both groups.

Advisor Insulin Guidance Software (Figure 1a) Subjects randomized to the experimental group received a PDA loaded with the insulin guidance software. At baseline (visit 1), a healthcare provider and/or certified diabetes educator (CDE) reviewed the features of the software on the PDA and loaded a subject specific insulin dosing algorithm into the software based on the physician's recommendations. The software program allowed the healthcare provider to enter demographic data such as age, height and weight which could potentially affect the insulin sensitivity factor already programmed into the device. The program advised basal, bolus and correction insulin dosages based on individual patients' prescriptions in addition to being alerted for SMBG testing. Subjects in the experimental group were also asked to input their blood glucose values into the PDA via the touch screen. Subjects then received a recommended insulin dose based on their prescription which was programmed by the healthcare provider. The patients were asked to either agree with the recommended insulin dose or disagree, and manually enter the insulin dose they took for a given event. All the data from the glucose meters and the PDAs were downloaded at every visit.

Glucose Target Ranges Glucose values were captured in one of the following categories to assess target glycemia and pie charts were created. Within Target Range (WTR) glucose values were those between 70-150mg/dL (3.89 to 8.33 mmol/L) (20). Below Target Range (BTR) glucose values were defined as ≤ 69mg/dL (3.83 mmol/L) and Above Target Range (ATR) glucose values were those values above 150mg/dL (8.33 mmol/L). These glucose levels were chosen based on our previous research on SMBG downloads (20).

Hypoglycemia Hypoglycemia was defined as glucose values ≤ 59mg/dL (3.27mmol/L). Severe hypoglycemia was defined as subjects needing assistance as previously described by DCCT Research Group (1).

A1c and Other Lab Measurement

The A1c values were measured by the DCA 2000® Analyzer, distributed by Bayer Corporation (Elkhart, IN). The DCA 2000® A1c assay gives accurate and precise results over a range of total hemoglobin from 7 to 24 g/dL. All subjects had hemoglobin concentrations well within these values. Normal A1c values are 3.4 to 6.2 % (18). The CBC (Beckman Coulter LH750, Beckman Coulter, Hialeah, FL), CMP (AU-5200 Olympus Japan Co Ltd, Tokyo) and CK (Olympus AU-800; Olympus, Tokyo, Japan) were performed by Quest Diagnostics, Denver, Colorado.

Statistical Analysis Wilcoxon Rank Sum and Chi Square tests of independence were used to compare continuous and categorical variables, respectively, at baseline. Chi Square test of independence was used to compare the number of discontinued subjects between the two groups. Mixed model repeated measures analysis with an unstructured covariance structure and pre-planned contrasts were used to compare the experimental and control groups on A1c, percent of glucose readings within, above, and below target, percent of total hypoglycemic events, basal insulin dose, weight, and BMI. Paired t-tests were used to test the within group change in weight from baseline to 12 months among those who completed all 12 months. Fisher's Exact test was used to compare the number of patients achieving target values between groups at each time point. Poisson regression was used to compare the frequency of severe hypoglycemic events between the two groups. Data are presented as least squares mean ± SE unless otherwise noted. All analyses were performed using SAS 9.1. Results were considered significant at p < 0.05 using a two-sided alpha.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, 18 to 60 years of age
* Diagnosed with Type 1 diabetes mellitus at least six months
* HbA1c 7.5% and 11.0% at screening
* Insulin dose 0.5 - 2.0 units/kg
* Hematocrit between 25% and 65%
* Weight 100-300 pounds
* On a dual insulin therapy supported by Accu-Chek Insulin Advisor software
* On a "day shift" schedule (typical day begins before noon)
* Willing to perform a minimum of three blood glucose tests per day - before breakfast, before lunch, and before dinner (standard of care)
* Willing to complete at least 7 clinic visits in 12 months (Baseline, 2-Week, 6-Week, 3-Month, 6-Month, 9-Month, and 12-Month)
* Willing to complete 3 study phone calls conducted by study coordinator (4.5-month, 7.5-Month and 10.5-Month)
* Able and willing to provide written informed consent to participate
* Willing to comply with the study protocol
* Willing to be randomized into either the Control Group or the Experimental Group

Exclusion Criteria:

* On insulin pump therapy
* On oral, inhaled or pre-mixed insulin
* Engaged in a minimum of 30 minutes of cardiovascular (aerobic) exercise 5 days out of a 7-day week
* Conditions that can cause significant increase of the insulin sensitivity factor, such as a steroid therapy, diabetic ketosis, insulin-resistant syndrome
* Creatinine above 2.5mg/dl, renal transplantation or currently undergoing kidney dialysis
* Pregnant or intends to become pregnant during the course of the study
* Undergoing therapy for a malignancy, other than basal cell or squamous cell skin cancer
* Plan to travel to a different time zone more than three times per month
* Clinical signs or symptoms of liver disease such as jaundice
* Diagnosis of acute or chronic hepatitis
* Diagnosis of hemoglobinopathy or chronic anemia
* Severe unexplained hypoglycemia in the past 3 months that required ED admission
* Participation in another clinical trial in the past 1 month
* Weight under 100 pounds or over 300 pounds

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 123 adult subjects ages 18-60 with type 1 diabetes on mulitiple daily injections
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2005-07; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Decrease in A1c of at least 0.4% in the insulin guidance software group as compared to the control group at 6 months and/or 1 year. | 1 year

SECONDARY OUTCOMES:
Hypoglycemic episodes, weight gain, insulin dose, frequency of self monitoring of glucose | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Satish K Garg, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Barbara Davis Center for Diabetes, Aurora, Colorado, United States